CLINICAL TRIAL: NCT06048081
Title: A Global, Multicenter, Open-label, Early Access Program for Zolbetuximab (IMAB362) Plus mFOLFOX6 or CAPOX in Patients With Claudin18.2-Positive, HER2-Negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Early Access Program for Zolbetuximab
Status: Available | Type: Expanded Access
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 8951-CL-9100
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Unresectable Gastroesophageal Junction (GEJ) Adenocarcinoma Cancer; Locally Advanced Unresectable Gastric Adenocarcinoma Cancer; Metastatic Gastric Adenocarcinoma Cancer; Metastatic Gastroesophageal Junction (GEJ) Adenocarcinoma
Keywords: Zolbetuximab; IMAB362; Modified oxaliplatin, folinic acid (leucovorin) and fluorouracim (FOLFOX6); Capecitabine and oxaliplatin (CAPOX); Early Access Program (EAP); Human epidermal growth factor receptor 2 (HER2) Negative; Claudin 18.2
MeSH Terms: conditions — Adenocarcinoma | interventions — zolbetuximab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: zolbetuximab — intravenous infusion
  mFOLFOX6 or CAPOX (used at physician discretion) will be used in combination with zolbetuximab
  Other Names: IMAB362

SUMMARY:
This program is to provide zolbetuximab to people with stomach cancer or gastroesophageal junction (the junction between stomach and esophagus) cancer who have not yet been treated with chemotherapy, immunotherapy, or zolbetuximab and who have tested positive for claudin18.2 (a protein found in some cancer cells). People will work with their doctor to see if they are capable of being treated with zolbetuximab while they receive other standard medicines to treat their cancer. The program will allow people early access to zolbetuximab before the drug is fully approved.

Zolbetuximab will be given through a vein. This is called an infusion. The infusion will happen during a person's treatment with other cancer medicines. Zolbetuximab will be given every 3 weeks. People will continue treatment until: they have medical problems (unwanted side effects) from the treatment; their cancer gets worse; they start other cancer treatment; they ask to stop treatment; or they do not come back for treatment.

People will visit the clinic on certain days during their treatment. During these visits, the program doctors will check for any medical problems (unwanted side effects) from zolbetuximab, other cancer treatment, or both. At some visits, other checks will include a medical examination, laboratory tests and vital signs. Vital signs include temperature, pulse, and blood pressure. Also, blood samples will be taken.

People will visit the clinic within 7 days after stopping treatment. The program doctors will check for any medical problems (unwanted side effects) from zolbetuximab or their cancer treatment. Other checks will include a medical examination, laboratory tests, and vital signs. Then, people will have a follow-up visit about 30 days after stopping treatment. If people are having no health problems, the follow-up visit can happen over the telephone.

DETAILED DESCRIPTION:
The European Union European Medicines Agency, the United States Food and Drug Administration, and South Korea Pharmaceuticals and Medical Devices Agency have approved zolbetuximab for the treatment of advanced stomach/GEJ cancer in adults. Enrollment is closed in United States, and Germany.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma.
* Patient has confirmed locally advanced, unresectable or metastatic gastric or GEJ adenocarcinoma.
* Patient whose tumor expresses claudin18.2 (CLDN18.2) in ≥ 75% of tumor cells demonstrating moderate to strong membranous CLDN18 staining as determined by local or central immunohistochemistry (IHC) testing.
* Patient has a Human epidermal growth factor receptor 2 (HER2-negative) tumor by local testing on a gastric or GEJ tumor specimen.
* Patient has Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patient must meet all of the following criteria based on the locally analyzed laboratory tests collected.

  * Hemoglobin (Hgb) ≥ 9 g/dL. Patients requiring transfusions are eligible if they have post-transfusion Hgb ≥ 9 g/dL.
  * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
  * Platelets ≥ 100 × 109/L
  * Albumin ≥ 2.5 g/dL
  * Total bilirubin (TBL) ≤ 1.5 × ULN without liver metastases (or < 3.0 × ULN if liver metastases are present)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN) without liver metastases (or ≤ 5 × ULN if liver metastases are present)
  * Estimated creatinine clearance ≥ 30 mL/min
  * Prothrombin time/international normalized ratio (PT/INR) and partial thromboplastin time ≤ 1.5 × ULN (except for patients receiving anticoagulation therapy)
* Female patient is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of child bearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 9 months after the final administration of oxaliplatin and 6 months after final administration of other interventions.
* Female patient must agree not to breastfeed starting at screening and throughout the EAP period and for 6 months after final intervention administration.
* Female patient must not donate ova starting at first administration of treatment and throughout the EAP period and for 9 months after the final administration of oxaliplatin and 6 months after final administration of other interventions.
* Male patient with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 6 months after final treatment administration.
* Male patient must not donate sperm during the treatment period and for 6 months after final treatment administration.
* Male patient with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the EAP period and for 6 months after final treatment administration.

Exclusion Criteria:

* Patient has previously received treatment in a clinical trial of zolbetuximab, or a clinical trial that included zolbetuximab as 1 of the treatment options, even if the patient was not given zolbetuximab.
* Patient is a candidate for an ongoing clinical trial of zolbetuximab.
* Patient has received any investigational therapy within 28 days or 5 half-lives prior to screening.
* Patient has a known or suspected hypersensitivity to zolbetuximab, other monoclonal antibodies or any components of the formulation used.
* Patient has received prior systemic chemotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma. However, patient may have received either neo-adjuvant or adjuvant chemotherapy, immunotherapy or other systemic anticancer therapies as long as it was completed at least 6 months prior to participation.
* Patient has received radiotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma ≤ 14 days prior to program registration and has not recovered from any related toxicity.
* Patient receiving treatment with herbal medications that have known antitumor activity.
* Patient has received systemic immunosuppressive therapy, including systemic corticosteroids within 14 days prior to registration. Patients using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg/day of hydrocortisone or up to 10 mg/day of prednisone), receiving a single dose of systemic corticosteroids or receiving systemic corticosteroids as premedication for radiologic imaging contrast use are allowed.
* Patient has a prior severe allergic reaction, known (immediate or delayed) or suspected hypersensitivity, intolerance or contraindication to zolbetuximab, mFOLFOX6, CAPOX, other monoclonal antibodies or any components of the formulations used.
* Patient has known dihydropyrimidine dehydrogenase (DPD) deficiency. (NOTE: Screening for DPD deficiency should be conducted per local requirements.)
* Patient has a complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent/recurrent vomiting.
* Patient has significant gastric bleeding and/or untreated gastric ulcers that would exclude the patient from participation.
* Patient has any other condition, which makes the patient unsuitable to receive or tolerate zolbetuximab.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (140):
- Site US10001, Morristown, New Jersey, United States
- Brazil (10):
  - BR55009, Belém
  - BR55001, Belo Horizonte
  - BR55004, Brasília
  - BR55002, Florianópolis
  - BR55007, Londrina
  - BR55010, Manaus
  - BR55008, Natal
  - BR55005, Porto Alegre
  - BR55003, Rio de Janeiro
  - BR55006, São Paulo
- France (86):
  - FR33004, Angers
  - FR33010, Angers
  - FR33054, Aubagne
  - FR33028, Avignon
  - FR33042, Bayeux
  - FR33040, Bobigny
  - FR33007, Bordeaux
  - FR33015, Bordeaux
  - FR33025, Brest
  - FR33046, Brieuc
  - FR33074, Brive-la-Gaillarde
  - FR33062, Caen
  - FR33021, Cagnes-sur-Mer
  - FR33073, Cagnes-sur-Mer
  - FR33086, Cholet
  - FR33013, Clermont-Ferrand
  - FR33024, Clermont-Ferrand
  - FR33026, Colmar
  - FR33065, Compiègne
  - FR33029, Corbeil-Essonnes
  - FR33083, Creil
  - FR33061, Créteil
  - FR33069, Dechy
  - FR33053, Gregoire
  - FR33039, Grenoble
  - FR33064, La Rochelle
  - FR33020, Le Blanc-Mesnil
  - FR33043, Lille
  - FR33084, Limoges
  - FR33063, Loches
  - FR33014, Lormont
  - FR33003, Lyon
  - FR33031, Lyon
  - FR33050, Mantes-la-Jolie
  - FR33001, Marseille
  - FR33045, Marseille
  - FR33008, Montpellier
  - FR33075, Montpellier
  - FR33049, Morlaix
  - FR33047, Moulins
  - FR33032, Nantes
  - FR33078, Nice
  - FR33035, Niort
  - FR33006, Paris
  - FR33011, Paris
  - FR33017, Paris
  - FR33033, Paris
  - FR33034, Paris
  - FR33080, Pau
  - FR33022, Perpignan
  - FR33012, Périgueux
  - FR33068, Plérin
  - FR33038, Poitiers
  - FR33048, Quincy-sous-Sénart
  - FR33058, Reims
  - FR33076, Rennes
  - FR33016, Rodez
  - FR33037, Rouen
  - FR33081, Rouen
  - FR33059, Saint-Etienne
  - FR33023, Saint-Grégoire
  - FR33079, Saint-Jean-de-Verges
  - FR33085, Saint-Martin-d'Hères
  - FR33056, Saint-Nazaire
  - FR33066, Saint-Priest-en-Jarez
  - FR33082, Saint-Priest-en-Jarez
  - FR33067, Saint-Quentin
  - FR33060, Sallanches
  - FR33071, Salon-de-Provence
  - FR33018, St-Malo
  - FR33005, Suresnes
  - FR33009, Suresnes
  - FR33057, Suresnes
  - FR33072, Thonon-les-Bains
  - FR33044, Tourcoing
  - FR33041, Tours
  - FR33055, Tours
  - FR33036, Trévenans
  - FR33070, Troyes
  - FR33051, Valenciennes
  - FR33002, Vannes
  - FR33030, Vantoux
  - FR33077, Verdun
  - FR33019, Villejuif
  - FR33027, Villejuif
  - FR33052, Villejuif
- Germany (26):
  - DE49020, Berlin
  - DE49021, Chemnitz
  - DE49004, Damme
  - DE49034, Damme
  - DE49006, Erkelenz
  - DE49030, Erkelenz
  - DE49029, Essen
  - DE49018, Frankfurt
  - DE49017, Frankfurt am Main
  - DE49003, Göttingen
  - DE49007, Hamburg
  - DE49033, Hamburg
  - DE49022, Kempten
  - DE49008, Kiel
  - DE49024, Kiel
  - DE49023, Koblenz
  - DE49019, Magdeburg
  - DE49010, Munich
  - DE 49005, München
  - DE49012, Nuremberg
  - DE49025, Ravensburg
  - DE49032, Thuine
  - DE49001, Tübingen
  - DE49002, Ulm
  - DE49011, Viersen
  - DE49016, Wiesbaden
- Singapore (6):
  - SG65001, Singapore
  - SG65002, Singapore
  - SG65003, Singapore
  - SG65004, Singapore
  - SG65005, Singapore
  - SG65006, Singapore
- South Korea (11):
  - KR82004, Incheon
  - KR82008, Seongnam-si
  - KR82001, Seoul
  - KR82002, Seoul
  - KR82003, Seoul
  - KR82006, Seoul
  - KR82007, Seoul
  - KR82009, Suwon
  - KR82010, Suwon
  - KR82011, Ulsan
  - KR82005, Yangsan